CLINICAL TRIAL: NCT03880110
Title: Combination of Biomarkers, Urine Sedimentation and Renal Resistive Index for Early Prediction of Acute Kidney Injury in High Risk Patients After Non-cardiac Surgery: a Prospective Observational Cohort Study
Brief Title: Early Prediction of Acute Kidney Injury in High Risk Patients After Non-cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Principal Investigator, Clinical Professor, Peking University First Hospital
Other Study IDs: Early predicting AKI
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Early prediction; Non cardiac surgery; Biomarker; Urine sedimentation; Renal resistive index
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After enrollment, blood and urine samples, in addition to clinical routine tests, will be collected for the tests of biomarkers and urine sedimentation, such as serum creatinine, TIMP-2, IGFBP-7, α-1 microglobulin, microalbumin, transferrin, granular cast and so on. Urine samples will be collected again for storage after 6 and 12 hours admitting to SICU, at which time urine sedimentation will be repeatedly measured at the discretion of physician in-charge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is a common complication after non-cardiac surgery with adverse short and long term morbidity and mortality. So far there have been no effective therapy for AKI treatment developed, possibly due to the heterogenicity of this syndrome. Therefore, prevention of AKI in high risk patients undergoing non-cardiac surgery, as emphasized by Kidney Disease Improving Global Outcomes (KDIGO), becomes the first priority. However, early prediction of AKI is the first step before taking preventive measures, which really make a great challenge to clinical practitioners because of such a limited time window and complex clinical scenarios. Recently, cumulative evidence have shown that biomarkers and renal ultrasound may play an important role in AKI prediction after non-cardiac surgery. The purpose of this study is to investigate the combination of biomarkers, urine sedimentation and renal resistive index for early prediction of AKI in high risk patients undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
Early prediction of AKI have long been a study hotspot. Various clinical prediction models, biomarkers, urine sedimentation scores and imaging tools are developed and validated in different clinical settings mainly focusing on contrast associated AKI, durg induced AKI and cardiac surgery associated AKI. Due to the heterogenicity of this syndrome, one parameter which fits all patients for prediction of AKI dose not possibly exist. As a result, searching for combination parameters that can well predict AKI after non-cardiac surgery become the first priority for prevention of AKI. Evidence in non-cardiac surgery population have been gradually accumulated in recent years. Biomarkers for G1 cell cycle arrest, e.g. tissue inhibitor of metalloproteinase-2 (TIMP-2) and insulin like growth factor binding protein-7 (IGFBP-7), have demonstrated robust predictive performance in high risk surgical patients. Renal resistive index as calculated by ultrasound have also showed its validity in AKI prediction in patients following orthopedic surgery. Hence, the investigators make an assumption that combination of biomarkers, urine sedimentation and renal resistive index may improve the predictive value of AKI after non-cardiac surgery. The purpose of this study is to investigate the combination of biomarkers, urine sedimentation and renal resistive index for early prediction of AKI in high risk patients undergoing non-cardiac surgery.

Adult patients undergoing non-cardiac surgery and then admitting to surgical intensive care unit (SICU) will be immediately screened for this study. After enrollment, blood and urine samples, in addition to clinical routine tests, will be collected for the tests of biomarkers and urine sedimentation, such as serum creatinine, TIMP-2, IGFBP-7, α-1 microglobulin, microalbumin, transferrin, granular cast and so on. Meanwhile, central venous pressure (CVP) will be measured by primary nurse. If the patients were enrolled at daytime between 8:00-16:00, experienced intensivists will also calculate the renal resistive index (RI) by ultrasound. Urine samples will be collected again for storage after 6 and 12 hours admitting to SICU, at which time urine sedimentation and CVP will be repeatedly measured at the discretion of physician in-charge. AKI is monitored by serum creatinine daily in SICU and on demand in general wards, and by urine output (UO) every 3 hours in SICU. Patients will be followed up for postoperative complications, renal recovery, survival, SICU/in hospital stay and total cost until the first thing that happens: discharge/death, 30d after operation or withdrawing the study. Perioperative data will be recorded by specialized researchers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; Undergoing non-cardiac surgery; Admitted to SICU immediately after surgery

Exclusion Criteria:

* Chronic kidney disease stage 5 (CKD-5) or requiring long-term dialysis; Undergoing kidney-related surgery; AKI before admission to SICU; Without Foley catheter placement ;Written informed consent not obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High risk patients undergoing non-cardiac surgery
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury within 7 days after surgery | within 7 days after surgery
  AKI is diagnosed according to KDIGO criteria

SECONDARY OUTCOMES:
Severity of acute kidney injury within 7 days after surgery | within 7 days after surgery
  AKI is classified according to KDIGO criteria
Incidence of postoperative complications | 30 days after operation or withdrawing the study ( the first thing that happens: discharge/death)
  Defined as newly onset medical conditions that are harmful to patients' recovery and required therapeutic intervention, including pulmonary infection, pleural effusion, atelectasis, respiratory failure, surgical bleeding, new onset arrhythmia, acute myocardial infarction, congestive heart failure, stroke, ileus, liver injury, digestive tract bleeding, wound infection, urinary tract infection, severe sepsis, acute kidney injury, pulmonary embolism and deep venous thrombosis.
Rate of ICU or in-hospital mortality | 30 days after operation or withdrawing the study ( the first thing that happens: discharge/death)
  ICU/In-hospital mortality
Rate of dialysis dependent at discharge | Until the first thing that happens: discharge/death, 30 days after operation or withdrawing the study.
  Defined as requiring any modality of renal replacement therapy at discharge
Rate of continuous decreased kidney function at discharge | 30 days after operation or withdrawing the study ( the first thing that happens: discharge/death)
  Estimated glomerular filtration rate (eGFR) decreased more than 25% of baseline value at discharge
Rate of major adverse kidney events (MAKE) | 30 days after operation or withdrawing the study ( the first thing that happens: discharge/death)
  Defined as a composite of death, dialysis dependent or continuous decreased kidney function

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grams ME, Sang Y, Coresh J, Ballew S, Matsushita K, Molnar MZ, Szabo Z, Kalantar-Zadeh K, Kovesdy CP. Acute Kidney Injury After Major Surgery: A Retrospective Analysis of Veterans Health Administration Data. Am J Kidney Dis. 2016 Jun;67(6):872-80. doi: 10.1053/j.ajkd.2015.07.022. Epub 2015 Sep 1. PMID 26337133
- [Background] Kashani K, Cheungpasitporn W, Ronco C. Biomarkers of acute kidney injury: the pathway from discovery to clinical adoption. Clin Chem Lab Med. 2017 Jul 26;55(8):1074-1089. doi: 10.1515/cclm-2016-0973. PMID 28076311
- [Background] Kashani K, Al-Khafaji A, Ardiles T, Artigas A, Bagshaw SM, Bell M, Bihorac A, Birkhahn R, Cely CM, Chawla LS, Davison DL, Feldkamp T, Forni LG, Gong MN, Gunnerson KJ, Haase M, Hackett J, Honore PM, Hoste EA, Joannes-Boyau O, Joannidis M, Kim P, Koyner JL, Laskowitz DT, Lissauer ME, Marx G, McCullough PA, Mullaney S, Ostermann M, Rimmele T, Shapiro NI, Shaw AD, Shi J, Sprague AM, Vincent JL, Vinsonneau C, Wagner L, Walker MG, Wilkerson RG, Zacharowski K, Kellum JA. Discovery and validation of cell cycle arrest biomarkers in human acute kidney injury. Crit Care. 2013 Feb 6;17(1):R25. doi: 10.1186/cc12503. PMID 23388612
- [Background] Bihorac A, Chawla LS, Shaw AD, Al-Khafaji A, Davison DL, Demuth GE, Fitzgerald R, Gong MN, Graham DD, Gunnerson K, Heung M, Jortani S, Kleerup E, Koyner JL, Krell K, Letourneau J, Lissauer M, Miner J, Nguyen HB, Ortega LM, Self WH, Sellman R, Shi J, Straseski J, Szalados JE, Wilber ST, Walker MG, Wilson J, Wunderink R, Zimmerman J, Kellum JA. Validation of cell-cycle arrest biomarkers for acute kidney injury using clinical adjudication. Am J Respir Crit Care Med. 2014 Apr 15;189(8):932-9. doi: 10.1164/rccm.201401-0077OC. PMID 24559465
- [Background] Gocze I, Koch M, Renner P, Zeman F, Graf BM, Dahlke MH, Nerlich M, Schlitt HJ, Kellum JA, Bein T. Urinary biomarkers TIMP-2 and IGFBP7 early predict acute kidney injury after major surgery. PLoS One. 2015 Mar 23;10(3):e0120863. doi: 10.1371/journal.pone.0120863. eCollection 2015. PMID 25798585
- [Background] Gunnerson KJ, Shaw AD, Chawla LS, Bihorac A, Al-Khafaji A, Kashani K, Lissauer M, Shi J, Walker MG, Kellum JA; Sapphire Topaz investigators. TIMP2*IGFBP7 biomarker panel accurately predicts acute kidney injury in high-risk surgical patients. J Trauma Acute Care Surg. 2016 Feb;80(2):243-9. doi: 10.1097/TA.0000000000000912. PMID 26816218
- [Background] Perazella MA. The urine sediment as a biomarker of kidney disease. Am J Kidney Dis. 2015 Nov;66(5):748-55. doi: 10.1053/j.ajkd.2015.02.342. Epub 2015 May 2. PMID 25943719
- [Background] Becker GJ, Garigali G, Fogazzi GB. Advances in Urine Microscopy. Am J Kidney Dis. 2016 Jun;67(6):954-64. doi: 10.1053/j.ajkd.2015.11.011. Epub 2016 Jan 22. PMID 26806004
- [Background] Marty P, Ferre F, Labaste F, Jacques L, Luzi A, Conil JM, Silva S, Minville V. The Doppler renal resistive index for early detection of acute kidney injury after hip fracture. Anaesth Crit Care Pain Med. 2016 Dec;35(6):377-382. doi: 10.1016/j.accpm.2015.12.013. Epub 2016 Apr 28. PMID 27133237
- [Background] Marty P, Szatjnic S, Ferre F, Conil JM, Mayeur N, Fourcade O, Silva S, Minville V. Doppler renal resistive index for early detection of acute kidney injury after major orthopaedic surgery: a prospective observational study. Eur J Anaesthesiol. 2015 Jan;32(1):37-43. doi: 10.1097/EJA.0000000000000120. PMID 25014511
- [Derived] Li N, Wang J, Zhou W, Li S, Yang L. External Validation of the Simple Postoperative Acute Kidney Injury Risk Index in Patients Admitted to the Intensive Care Unit After Noncardiac Surgery. Anesth Analg. 2025 May 1;140(5):1140-1148. doi: 10.1213/ANE.0000000000007320. PMID 39919018
- [Derived] Li N, Zhou WJ, Chi DX, Yuan C, Xie M, Li Z, Wang R, Qu CX, Li XY, Li SL, Yang L. Association between urine microscopy and severe acute kidney injury in critically ill patients following non-cardiac surgery: a prospective cohort study. Ann Palliat Med. 2022 Jul;11(7):2327-2337. doi: 10.21037/apm-21-3085. Epub 2022 May 19. PMID 35610195